CLINICAL TRIAL: NCT05736848
Title: A Retrospective Assessment of OviTex PRS (OviTex) Permanent and Resorbable Devices in Subjects Who Have Previously Undergone a Breast Reconstruction
Brief Title: A Retrospective Assessment of OviTex PRS (OviTex)
Acronym: PRS
Status: Recruiting | Type: Observational
Sponsor: Tela Bio Inc (Industry)
Collaborators: MCRA (Industry)
Responsible Party: Sponsor
Other Study IDs: TB2022.01.02
Record Dates: First submitted 2023-01-23; First posted 2023-02-21 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Reconstructive Surgical Procedures

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: OviTex® PRS — OviTex® PRS is a reinforced tissue matrix intended to reinforce soft tissue where weakness exists in patients requiring soft tissue repair or reinforcement in plastic and reconstructive surgery.
  Other Names: OviTex PRS Permanent - Pre-pectoral; OviTex PRS Permanent - Sub-pectoral; OviTex PRS Resorbable - Pre-pectoral; OviTex PRS Resorbable - Sub-pectoral

SUMMARY:
The objective of this retrospective-prospective, observational study is to evaluate the safety profile overall and within two device types of OviTex PRS in previous pre-pectoral or sub-pectoral implant-based breast reconstructions.

DETAILED DESCRIPTION:
This study is organized as a retrospective-prospective, observational, multi-center study. The treatment group involved in the study received OviTex PRS during implant-based breast reconstruction. The reconstruction procedure was an immediate or two-stage unilateral or bilateral implant in either the sub-pectoral or pre-pectoral position. Results from this study are aimed to demonstrate an acceptable safety profile and to inform the study design and effectiveness endpoints of a future prospective study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient was between 18 years and 75 years of age (inclusive) at the time of surgery.
2. At the time of surgery, the patient received an OviTex PRS Permanent (R20143 or R20243) or Resorbable (R20152 or R20252) implant in conjunction with an implant-based breast reconstruction.
3. Patient has undergone their initial surgical procedure and exchange surgery (if applicable).

Exclusion Criteria:

1. Patient received a textured permanent breast implant.
2. Patient was a nicotine user (including smokeless, vaporized, etc.) within 4-weeks preceeding their index procedure.
3. Patient had previously undergone radiation therapy to the chest wall prior to index surgery.

Additional prospective inclusion criteria (if applicable):

1. Patient agrees to return in-person for prospective portion including the completion of photographs.

Additional prospective exclusion criteria (if applicable):

1. Patient has a history of a psychological condision, drug or alcohol abuse which may interfere with their ability to adhere to the follow-up requirements.

Ages: 18 Years to 75 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Data will be collected for 200 subjects that have been implanted with OviTex® PRS
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2022-09-27 (Actual); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
The occurrence of relevant (S)AEs within 24 months of OviTex® PRS implantation. | 24 months
  Retrospective - Prospective assessment

SECONDARY OUTCOMES:
Time to Expander/Implant Exchange | 24-months
  Retrospective - Prospective assessment
Intraoperative Fill Volume / Number and Volume of Fill Visits | 24 months
  Retrospective - Prospective assessment
Independent aesthetic assessment of each treated breast as measured by Telemark Breast Score | 24 months
  Image aesthetic assessment
Independent assessment of breast ptosis as measured by the Rainbow Scale | 24-months
  Retrospective - Prospective assessment
Hospitalization length of stay | At procedure
  Retrospective - Prospective assessment

CONTACTS AND LOCATIONS:
Overall Officials: Asaf Yalif, MD, Principal Investigator — Y Plastic Surgery
Locations (11):
- United States (11):
  - Aesthetic Surgery Center, Naples, Florida
  - Castrellon Aesthetic Surgery, South Miami, Florida
  - Y Plastic Surgery, Alpharetta, Georgia
  - Massachusetts General Hospital, Boston, Massachusetts
  - Janineh Plastic Surgery, Rochester Hills, Michigan
  - David L. Abramson, MD, Englewood, New Jersey
  - Capital Health, Pennington, New Jersey
  - Strong Memorial Hospital, Rochester, New York
  - Plastic Surgery Consultants, Columbia, South Carolina
  - Dermatology Associates of San Antonio/Baptist Medical Center, San Antonio, Texas
  - Houston Methodist The Woodlands Hospital, The Woodlands, Texas

IPD SHARING:
Plan to Share IPD: No